CLINICAL TRIAL: NCT00712621
Title: Phase II Two Arm Randomized Controlled Clinical Trial to Study Quality of Life and Survival of Breast Cancer Patients After Completion of Chemotherapy or Radiation Therapy or Surgery or Any Combination Therapy in Stage I to IV Carcinoma
Brief Title: Determining Quality of Life in Breast Cancer Patient After Completing Radiation,Chemotherapy,Surgery or Combination
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is withdrawn due to unavailability of eligible subject population. We will request the sponsors to extend the time for enrollment.
Sponsor: American Scitech International (Other)
Responsible Party: Dr. Ratna Grewal, American Scitech International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ASI-QOLII0608; ASI-QOL8655
Record Dates: First submitted 2008-06-18; First posted 2008-07-10 (Estimated); Last update posted 2009-11-24 (Estimated); Status verified 2009-11

CONDITIONS: Breast Carcinoma
Keywords: Genetics Home Reference related topics; breast cancer; breast cancer related to depression; Condition; Stage I-IV Carcinoma of Breast
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Counseling; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Other): OUTLINE: This is a randomized, multicenter study. Patients are selected according to age ( 25 to 49 vs 50 to 85), time since initial completion of therapy (3 to 18 months), and are separated in two groups.
  Arm I: Quality of life is assessed at baseline and at 3 and 6 months.
  Interventions: Behavioral: Written materials
- II (Other): OUTLINE: This is a randomized, multicenter study. Patients are selected according to age ( 25 to 49 vs 50 to 85), time since initial completion of therapy (3 to 18 months), and are separated in two groups.
  Arm II: Quality of life is assessed at baseline and at 3 and 6 months.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — • Arm II: Patients receive audio visual aids and weekly counseling sessions by the expert counselors and breast cancer survivors over 8 weeks for a total of 8-16 sessions. Patients receive written materials from the counseling group after the completion of the sessions
  Other Names: Lifestyle Counseling
  Arms: II
Behavioral: Written materials — • Arm I: Patients receive the support by providing existing resources. Patients receive standard written materials from the counseling group after enrolling in the study.
  Other Names: Quality of Life
  Arms: I

SUMMARY:
Rationale: Determining quality of life in breast cancer patient after completing chemotherapy or radiation therapy or surgical procedures or any combination therapy.

Intervention includes supportive care in terms of psychological support and moral boosting efforts by counseling breast cancer survivors which may enhance the well-being and quality of life of women who are treated with chemotherapy or radiation therapy or surgical procedures or any given combination therapy.

PURPOSE: Randomized clinical trial study to compare the effectiveness of support system and counseling of breast cancer survivors on the well-being of women, who have completed various modes of treatment of breast cancer with the subjects who have no support system.

Study Type: Quality of life and survival

Study Design: Two arm randomized controlled clinical trial to study quality of life and survival of breast cancer patients after completion of chemotherapy or radiation therapy or surgery or any combination therapy. The stages from I to IV (metastases to other sites of the body) are included.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the quality of life in breast cancer patient after completing chemotherapy or radiation therapy or surgical procedures or any combination therapy in both Arms.
* Determine the effect of providing standard written materials in Arm I.
* Determine the effect of psychological support and moral boosting efforts by counseling breast cancer survivors which may enhance the well-being and quality of life of women who are treated with chemotherapy or radiation therapy or surgical procedures or any combination therapy in Arm II.
* Determine the effect of socioeconomic status on all available demographic area which is not a criteria for exclusion in both Arms.
* Determine psychosocial and mental state to measure wellness and good quality of life in both Arms.
* Determine the periodic medical care for related or unrelated problems of the disease which have a positive impact on the survival and quality of life in both Arms.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients
* 25 to 85 years old

DISEASE CHARACTERISTICS:

* Received prior definitive treatment for stage I-IV breast cancer with or without adjuvant chemotherapy or radiation therapy or surgical therapy or any combination therapy.
* 3 to 18 months since completion therapy.

PATIENT CHARACTERISTICS:

Age:

* 25 to 49 vs 50 to 85

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* CBC in normal range:
* Hemoglobin - 10 g/dl
* Blood Glucose is twofold above the normal range

Hepatic:

* Hepatic profile is twofold above the normal range:
* AST/ALT
* Bilirubin,total
* Protein (Albumin, Globulin)

Renal:

* Renal tests are twofold above the normal range:
* Creatinine clearance 24 hours
* BUN
* Creatinine level

Other:

* No current psychiatric diagnosis
* Mini Mental Status Examination
* No signs and symptoms MDD
* Anxiety disorder
* Post Traumatic Syndrome Disorder

Status of Therapy:

Chemotherapy:

* Completed

Endocrine therapy:

* Completed

Radiotherapy:

* Completed

Surgery:

* Completed at least three months before the start of the study

Exclusion Criteria:

* Age below 25 and above 85
* Subject with breast carcinoma in therapy
* Any current mental illness
* Hepatic enzymes are more than twofold from the normal range
* Renal impairment is more than twofold from the normal range
* Hemoglobin is less than 10 g/dl
* CBC results are below normal range

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2010-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Procedure: Psychological assessment and discussion on social & economic issues and medical problems related or unrelated to the therapy; quality-of-life assessment; long term survival | 2-4 years

SECONDARY OUTCOMES:
Long term disease free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Prem A Nandiwada, MD, Principal Investigator — Raritan Bay Medical Center; Ratna Grewal, MD, Study Chair — American Scitech International-eCRO; Sarat Babu, MD, Study Director — St. Peter's Hospital
Locations (1):
- Practicing physician in New Jersey, Englishtown, New Jersey, United States